CLINICAL TRIAL: NCT05976490
Title: NeuroPathways: An Information and Support Intervention for Patients With Malignant Brain Tumors
Brief Title: NeuroPathways Intervention for Brain Tumor Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Deborah A Forst, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-178
Record Dates: First submitted 2023-07-18; First posted 2023-08-04 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Malignant Brain Tumor; Glioma; Coping Skills
Keywords: glioma; supportive care; psychoeducation; information
MeSH Terms: conditions — Brain Neoplasms; Glioma

STUDY DESIGN:
Intervention Model Description: Open pilot to refine the intervention in up to 10 participants, followed by a pilot randomized controlled trial (n=40) in which participants will be randomized 1:1 to the intervention versus usual care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NeuroPathways Open Pilot (Experimental): Enrolled patients will receive an intervention guide with information about navigating life with a brain tumor diagnosis, and will participate in four weekly or biweekly, individual sessions with a clinician (e.g. nurse or behavioral health specialist).
  Participants will be asked to complete surveys at baseline, 8 weeks and 12 weeks, as well as an exit interview after the intervention.
  Interventions: Behavioral: Information and Support Intervention
- NeuroPathways Pilot RCT (Experimental): Enrolled patients will receive an intervention guide with information about navigating life with a brain tumor diagnosis, and will participate in four weekly or biweekly, individual sessions with a clinician (e.g. nurse or behavioral health specialist).
  Participants will be asked to complete surveys at baseline, 8 weeks and 12 weeks.
  Interventions: Behavioral: Information and Support Intervention
- Usual supportive care (Active Comparator): Participants will receive usual supportive care, which includes referral to cancer center supportive care services (e.g., social work) upon request from the patient, caregiver, or clinician.
  Participants will be asked to complete surveys at baseline, 8 weeks and 12 weeks.
  Interventions: Other: Usual supportive care

INTERVENTIONS:
Behavioral: Information and Support Intervention — Information guide and four one-on-one coaching sessions
  Other Names: NeuroPathways
  Arms: NeuroPathways Open Pilot; NeuroPathways Pilot RCT
Other: Usual supportive care — Referral to cancer center supportive care services (e.g., social work) upon request from the patient, caregiver, or clinician
  Arms: Usual supportive care

SUMMARY:
This goal of this study is to test an information and support intervention for patients with malignant (or "high-grade") brain tumors. This study was developed to help patients cope after a brain tumor diagnosis. The main question this study aims to answer is whether this intervention (which includes access to an information guide and one-on-one coaching sessions) is feasible (i.e., possible to carry out) and acceptable (i.e., considered helpful) to patients. Participants will be asked to take part in the coaching sessions, use the guide as desired, and complete a small group of short surveys at three different points in time; some participants will be asked to share feedback via exit interviews.

DETAILED DESCRIPTION:
This study will be a prospective pilot randomized controlled trial to examine the feasibility and acceptability of a novel, population-specific intervention designed to help patients with recently-diagnosed malignant brain tumors process and cope with their illness.

The specific aims are to 1) refine the NeuroPathways intervention based on feedback from an open pilot study (n=up to 10) with exit interviews, 2) evaluate the feasibility and acceptability of NeuroPathways in a pilot randomized controlled trial (n=40), and 3) explore preliminary effects of the intervention on psychological, behavioral, and cognitive outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Massachusetts General Hospital Cancer Center patient
* Within 6 weeks of diagnosis with a primary malignant brain tumor
* Able to speak and read in English

Exclusion Criteria:

* Inability to provide informed consent as assessed by the study team (e.g., due to neurological impairment such as severe cognitive impairment/dementia or moderate-to-severe receptive aphasia)
* Deemed inappropriate to approach by patient's oncologist or study PI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-11-07 (Actual); Primary Completion 2026-09-10 (Estimated); Study Completion 2027-04-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the Intervention: Percentage of Eligible Patients Who Enroll and Participate in the Intervention | 2 years
  The investigators will assess feasibility by examining the percentage of eligible patients who agree to enroll in the study and the percentage of enrolled patients who participate in all four intervention sessions. The intervention will be deemed feasible if at least 60% of eligible patients enroll in the study and if at least 60% of enrolled patients complete all four sessions.
Acceptability of the Intervention: Percentage of Participants who Have High Satisfaction with the Intervention | 2 years
  The investigators will assess acceptability via examining the distribution of patient scores for the 8-item Client Satisfaction Questionnaire (CSQ-8). CSQ-8 scores range from 8 to 32, with higher scores indicating higher satisfaction. The intervention will be deemed acceptable if at least 80% of patients score at least 20 points on the CSQ-8.

OTHER OUTCOMES:
Exploratory: Perceived Cognitive Function | 2 years
  The investigators will explore the effect of NeuroPathways on perceived cognitive function using the Functional Assessment of Cancer Therapy - Cognitive Function (FACT-Cog) between study arms in the pilot RCT phase of this study. The FACT-Cog is a 37-item measure of perceived cognitive impairment in cancer patients with scores from 0-148 and higher scores representing higher perceived cognitive functioning.
Exploratory: Distress (Depression and Anxiety Symptoms) | 2 years
  The investigators will explore the effect of NeuroPathways on distress using the Hospital Anxiety and Depression Scale (HADS) between study arms in the pilot RCT phase of this study. The HADS is a 14-item questionnaire that contains two 7-item subscales assessing depression and anxiety symptoms during the past week. Used extensively in samples of patients with cancer and their caregivers, the questionnaire consists of a four-point item response format that quantifies the degree to which participants experience mood symptoms. Scores on each subscale range from 0 to 21, with higher scores indicating higher symptom burden, and a cutoff of 8 or greater denoting clinically significant anxiety or depression.
Exploratory: Self-Efficacy | 2 years
  The investigators will explore the effect of NeuroPathways on self-efficacy using the Lewis Cancer Self-Efficacy Scale (CASE) between study arms in the pilot RCT phase of this study. The CASE is a 17-item questionnaire with a score range of 0-170. Higher scores reflect higher confidence in managing the impact of one's illness.
Exploratory: Loneliness | 2 years
  The investigators will explore the effect of NeuroPathways on loneliness using the Patient-Reported Outcomes Measurement Information System (PROMIS) - Social Isolation between study arms in the pilot RCT phase of this study. The PROMIS - Social Isolation is a 8-item questionnaire, scored from 4-20, that is used to evaluate feelings of loneliness and social isolation. Higher scores indicate greater feelings of loneliness and social isolation.
Exploratory: Coping | 2 years
  The investigators will explore the effect of NeuroPathways on coping using the Brief Coping Orientation to Problems Experienced (Brief-COPE). The Brief-COPE is a 28-item self-report measure assessing a variety of coping styles with scores ranging from 28-112 and higher scores indicating greater coping ability.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah A Forst, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to the principal investigator, Deborah Forst, MD.
  The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Time Frame: Data can be shared no earlier than 1 year following the date of publication.
Access Criteria: Only de-identified participant data from the final research dataset used in the published manuscript can be shared. Data shall only be shared upon request with researchers who provide a methodologically sound research proposal, at the discretion of the principal investigator.